CLINICAL TRIAL: NCT06191250
Title: Short Pre-sUrgical Plan in Locally Advanced Non-small Cell Lung Cancer Employing Radiation, Immuno-Oncology and Resection
Brief Title: --SuPERIOR Trial--
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study Terminated Prior to trial activation, due to changes in SOC of the treatment
Sponsor: University Health Network, Toronto (Other)
Collaborators: Ontario Institute for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SuPERIOR
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC); Clinical Staging T2b-3 N0-1 M0
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab

STUDY DESIGN:
Intervention Model Description: This is a multi-centre, phase 2, WOO trial in patients with T2b-3N0-1M0 NSCLC evaluating the biologic efficacy of NORT-durvalumab administered prior to surgery. The trial will assess the feasibility of the study design using neoadjuvant NORT-durvalumab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant NORT-durvalumab (Experimental): administration of non-ablative oligofractionated radiation therapy using 12 Gy in 3 fractions in combination with one dose of durvalumab (750 mg IV) prior to surgery.
  Interventions: Drug: Durvalumab; Radiation: Non-ablative oligofractionated radiation (NORT)

INTERVENTIONS:
Drug: Durvalumab — one dose of durvalumab (750 mg IV)
Radiation: Non-ablative oligofractionated radiation (NORT) — 12 Gy of Radiation in 3 fractions

SUMMARY:
The Window-of-Opportunity (WOO) Network is a collaboration among Ontario's doctors and scientists to conduct clinical trials in newly-diagnosed cancer patients before they have surgery with an initial focus on understanding how cancer drugs can impact the immune system.

There is often a waiting period of two to six weeks between when a patient first receives a cancer diagnosis and their scheduled surgery. This period provides a unique opportunity to study tumours before they are treated, allowing scientists to explore new ways to identify cancer, measure how cancer cells respond to treatment, and understand how therapies work. WOO Network trials include drugs or treatments that already have been tested in other clinical trials or are already approved by Health Canada.

The SuPERIOR trial is a WOO trial and it is designed for cohort of patients patients diagnosed with newly-diagnosed cancer patients with stage two or three non-small cell lung cancer.

The patients who are enrolled in this trial will received combination of Non-ablative oligofractionated radiation (NORT) which is a low dose of radiation and one dose of Durvalumab, an immunotherapy drug before their surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of study entry.
2. Written informed consent.
3. Pathologically proven NSCLC irrespective of PD-L1 expression status.
4. Tumor tissue is available for the mandatory translational research.
5. Tumor stage T2b-3N0-1M0 according to the TNM classification, 8th edition.
6. Tumor is considered resectable.
7. ECOG performance status 0-1.
8. Adequate hematological values: hemoglobin ≥ 90 g/L, absolute neutrophils count ≥ 1.5 x 109/L, platelets count ≥ 100 x 109/L.
9. Adequate hepatic function: bilirubin ≤ 1.5 x ULN, AST/ALT ≤ 1.5 x ULN, AP ≤ 2.5 x ULN.
10. Adequate renal function: calculated creatinine clearance ≥ 60 mL/min, according to the formula of Cockcroft-Gault.
11. Women with child-bearing potential who are using effective contraception, are not pregnant or lactating and agree not to become pregnant during participation in the trial and during 90 days after the last treatment. A negative serum pregnancy test performed within 7 days before registration into the trial is required for all women with child-bearing potential. Men agree not to father a child during participation in the trial and during 90 days after the last treatment.
12. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow-up.

Exclusion Criteria:

1. Presence of any distant metastasis or N2 or N3 disease.
2. Patients with a history of other malignancies, except non-active malignancy that does not require treatment, nor anticipated to require treatment for the duration of the study, and in the opinion of the investigator would not pose a risk of increased toxicity, or difficulty to follow the protocol and assess endpoints of the study.
3. Any previous treatment with a PD-1 or PD-L1 inhibitor, including durvalumab.
4. Absolute contraindications for the use of corticosteroids as premedication.
5. Concurrent treatment with other experimental drugs or other anti-cancer therapy, treatment in a clinical trial within 30 days prior to registration.
6. Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses (i.e., which must not exceed 10 mg/day of prednisone or an equivalent corticosteroid).
7. Severe or uncontrolled cardiac disease requiring treatment, congestive heart failure NYHA III or IV, unstable angina pectoris even if medically controlled, history of myocardial infarction during the last 3 months, serious arrhythmias requiring medication (with exception of atrial fibrillation or paroxysmal supraventricular tachycardia).
8. Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Bazett's Correction.
9. Body weight less than 30 kg.
10. Active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease or a syndrome that requires systemic steroids or immunosuppressive agents. Exceptions: - Vitiligo or resolved childhood asthma/atopy - Hypothyroidism stable on hormone replacement or Sjorgen's syndrome
11. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
12. Known evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection.
13. History of primary immunodeficiency.
14. History of allogeneic organ transplant.
15. Receipt of live attenuated vaccination within 30 days prior to the first dose of durvalumab (COVID-19 vaccine is permitted).
16. Any concomitant drugs contraindicated for use with durvalumab: this includes systemic corticosteroids, methotrexate, azathioprine, and tumor necrosis factor (TNF)-α blockers. Any concomitant drugs contraindicated for use with the other trial drugs according to the locally approved product information.
17. Any other serious underlying medical (e.g., uncontrolled diabetes mellitus, active uncontrolled infection, active gastric ulcer, uncontrolled seizures, severe hearing impairment), psychiatric, psychological, familial or geographical condition that, in the judgment of the investigator, may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-09-28 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Measuring CD8 TILs density post NORT-durvalumab | 17 days
  Neoadjuvant durvalumab in combination with non-ablative oligofractionated radiation therapy (NORT) using 12 Gy in 3 fractions can upregulate CD8+ tumor infiltrating lymphocytes (TILs) in T2b-3 N0-1 M0 non-small cell lung cancer (NSCLC)

CONTACTS AND LOCATIONS:
Overall Officials: Marc de Perrot, MD, MSc, FRCSC, Principal Investigator — Toronto General Hospital
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No